CLINICAL TRIAL: NCT06311214
Title: Optimizing Antibody-Drug Conjugate Therapy Through Molecular Analysis for Therapy Choice (ADC MATCH)
Brief Title: Personalized Antibody-Drug Conjugate Therapy Based on RNA and Protein Testing for the Treatment of Advanced or Metastatic Solid Tumors (The ADC MATCH Screening and Treatment Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01903; NCI-2024-01903 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10397 (Other: University of Texas MD Anderson Cancer Center LAO); 10397 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2024-03-13; First posted 2024-03-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; enfortumab vedotin; Immunohistochemistry; Magnetic Resonance Spectroscopy; sacituzumab govitecan; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A (sacituzumab govitecan) (Experimental): Patients receive sacituzumab govitecan IV over 1-3 hours on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the trial, undergo biopsy after enrollment to cohort but prior to treatment and again on study, and undergo collection of blood samples after enrollment to cohort but prior to treatment. Patients may optionally undergo biopsy at the time of progression and may optionally undergo collection of blood samples on study and at the time of progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Sacituzumab Govitecan
- Cohort B (enfortumab vedotin) (Experimental): Patients receive enfortumab vedotin IV over 30 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the trial, undergo biopsy after enrollment to cohort but prior to treatment and again on study, and undergo collection of blood samples after enrollment to cohort but prior to treatment. Patients may optionally undergo biopsy at the time of progression and may optionally undergo collection of blood samples on study and at the time of progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Enfortumab Vedotin; Procedure: Magnetic Resonance Imaging
- Cohort C (trastuzumab deruxtecan) (Experimental): Patients receive trastuzumab deruxtecan IV over 90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the trial, undergo biopsy after enrollment to cohort but prior to treatment and again on study, and undergo collection of blood samples after enrollment to cohort but prior to treatment. Patients also undergo ECHO or MUGA at screening and on study. Patients may optionally undergo biopsy at the time of progression and may optionally undergo collection of blood samples on study and at the time of progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Trastuzumab Deruxtecan
- Screening (record review, IHC assay) (Other): SCREENING STEP 1: Patients who have previously undergone SOC RNA testing have the results of their SOC RNA testing reviewed. Patients whose tumor expresses an appropriate TOI by RNA testing proceed to screening step 2.
  SCREENING STEP 2: Patients have TOI expression testing at the protein level by IHC assay performed on previously collected tissue. Patients with high Trop-2 protein expression are assigned to Cohort A. Patients with high nectin-4 protein expression are assigned to Cohort B. Patients with high HER2 protein expression are assigned to cohort C.
  Interventions: Other: Electronic Health Record Review; Other: Immunohistochemistry Staining Method

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Cohort A (sacituzumab govitecan); Cohort B (enfortumab vedotin); Cohort C (trastuzumab deruxtecan)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Cohort A (sacituzumab govitecan); Cohort B (enfortumab vedotin); Cohort C (trastuzumab deruxtecan)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Cohort A (sacituzumab govitecan); Cohort B (enfortumab vedotin); Cohort C (trastuzumab deruxtecan)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: Cohort C (trastuzumab deruxtecan)
Other: Electronic Health Record Review — Undergo review of SOC RNA testing results
  Arms: Screening (record review, IHC assay)
Drug: Enfortumab Vedotin — Given IV
  Other Names: AGS 22ME; AGS-22M6E; Anti-Nectin 4 ADC ASG-22CE; Anti-nectin-4 Monoclonal Antibody-Drug Conjugate AGS-22M6E; ASG 22CE; ASG-22CE; ASG22CE; Enfortumab Vedotin-ejfv; Padcev
  Arms: Cohort B (enfortumab vedotin)
Other: Immunohistochemistry Staining Method — Undergo IHC assay
  Other Names: Cell/Tissue, Immunohistochemistry; IHC; Immunohistochemistry; Immunohistochemistry (IHC)
  Arms: Screening (record review, IHC assay)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Cohort A (sacituzumab govitecan); Cohort B (enfortumab vedotin); Cohort C (trastuzumab deruxtecan)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Cohort C (trastuzumab deruxtecan)
Biological: Sacituzumab Govitecan — Given IV
  Other Names: hRS7-SN38 Antibody Drug Conjugate; IMMU 132; IMMU-132; IMMU132; RS7 SN38; RS7-SN38; RS7SN38; Sacituzumab Govitecan-hziy; Trodelvy
  Arms: Cohort A (sacituzumab govitecan)
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; T-DXd; WHO 10516
  Arms: Cohort C (trastuzumab deruxtecan)

SUMMARY:
This phase II ADC MATCH screening and multi-sub-study treatment trial is evaluating whether biomarker-directed treatment with one of three antibody-drug conjugates (ADCs) (sacituzumab govitecan, enfortumab vedotin, and trastuzumab deruxtecan) works in treating patients with solid tumor cancers that have high expression of the Trop-2, nectin-4, or HER2 proteins and that may have spread from where they first started (primary site) to nearby tissue, lymph nodes, or distant parts of the body (advanced) or to other places in the body (metastatic). Precision medicine is a form of medicine that uses information about a person's genes, proteins, and environment to prevent, diagnose, or treat disease in a way that is tailored to the patient. ADCs such as sacituzumab govitecan, enfortumab vedotin, and trastuzumab deruxtecan are monoclonal antibodies attached to biologically active drugs and are a form of targeted therapy. Sacituzumab govitecan is a monoclonal antibody, called sacituzumab, linked to a drug called govitecan. Sacituzumab attaches to a protein called Trop-2 on the surface of tumor cells and delivers govitecan to kill them. Enfortumab vedotin is a monoclonal antibody, enfortumab, linked to an anticancer drug called vedotin. It works by helping the immune system to slow or stop the growth of tumor cells. Enfortumab attaches to a protein called nectin-4 on tumor cells in a targeted way and delivers vedotin to kill them. Trastuzumab deruxtecan is composed of a monoclonal antibody, called trastuzumab, linked to a chemotherapy drug, called deruxtecan. Trastuzumab attaches to HER2 positive tumor cells in a targeted way and delivers deruxtecan to kill them. Personalized treatment with sacituzumab govitecan, enfortumab vedotin, or trastuzumab deruxtecan may be an effective treatment option for patients with advanced or metastatic solid tumors that screen positive for high expression of Trop-2, nectin-4, or HER2, respectively.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the proportion of patients with expression of targets of interest (TOIs) by ribonucleic acid (RNA) testing who have expression of the TOI protein by immunohistochemistry (IHC). (ADC MATCH screening protocol) II. To evaluate the objective response rate (ORR) of patients with advanced/metastatic solid tumors and high TOI protein expression to matched ADCs. (ADC MATCH treatment cohorts)

SECONDARY OBJECTIVES:

I. To determine the proportion of patients with high validated TOI protein expression who receive treatment on ADC MATCH. (ADC MATCH screening protocol) II. To evaluate the proportion of patients with advanced/metastatic solid tumors who are alive and progression free at 6 months of treatment with targeted ADC. (ADC MATCH treatment cohorts) III. To evaluate time until death or disease progression. (ADC MATCH treatment cohorts) IV. To determine progression-free survival (PFS) compared to prior line of therapy (PFS2/PFS1). (ADC MATCH treatment cohorts) V. To determine the correlation of RNA and protein expression of TOIs. (ADC MATCH treatment cohorts) VI. To determine temporal tumor heterogeneity by comparing RNA/protein expression of TOIs on archival samples versus fresh biopsies. (ADC MATCH treatment cohorts) VII. To identify potential predictive biomarkers, including target expression (RNA and protein) and other molecular features (deoxyribonucleic acid [DNA], RNA, protein, immune markers). (ADC MATCH treatment cohorts) VIII. To determine pharmacodynamic changes in the tumor and microenvironment. (ADC MATCH treatment cohorts)

EXPLORATORY OBJECTIVE:

I. To determine mechanisms of acquired resistance. (ADC MATCH treatment cohort)

OUTLINE:

SCREENING STEP 1: Patients who have previously undergone standard of care (SOC) RNA testing have the results of their SOC RNA testing reviewed. Patients whose tumor expresses an appropriate TOI by RNA testing proceed to screening step 2.

SCREENING STEP 2: Patients have TOI expression testing at the protein level by IHC assay performed on previously collected tissue. Patients with high Trop-2 protein expression are assigned to Cohort A. Patients with high nectin-4 protein expression are assigned to Cohort B. Patients with high HER2 protein expression are assigned to cohort C.

COHORT A: Patients receive sacituzumab govitecan intravenously (IV) over 1-3 hours on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) throughout the trial, undergo biopsy after enrollment to cohort but prior to treatment and again on study, and undergo collection of blood samples after enrollment to cohort but prior to treatment. Patients may optionally undergo biopsy at the time of progression and may optionally undergo collection of blood samples on study and at the time of progression.

COHORT B: Patients receive enfortumab vedotin IV over 30 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the trial, undergo biopsy after enrollment to cohort but prior to treatment and again on study, and undergo collection of blood samples after enrollment to cohort but prior to treatment. Patients may optionally undergo biopsy at the time of progression and may optionally undergo collection of blood samples on study and at the time of progression.

COHORT C: Patients receive trastuzumab deruxtecan IV over 90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the trial, undergo biopsy after enrollment to cohort but prior to treatment and again on study, and undergo collection of blood samples after enrollment to cohort but prior to treatment. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) at screening and on study. Patients may optionally undergo biopsy at the time of progression and may optionally undergo collection of blood samples on study and at the time of progression.

At the time that a confirmed objective response is observed for a specific tumor type in any cohort, that tumor type may be expanded into a separate tumor-specific expansion cohort, with up to 2 expansion cohorts allowed per treatment cohort. At the time of disease progression, patients with expression of additional TOIs may be re-screened and assigned to receive treatment in up to 2 of the other treatment cohorts.

After completion of study treatment, patients are followed up at 30 days then every 3 months in years 1-2 and every 6 months in year 3.

ELIGIBILITY:
Inclusion Criteria:

* SCREENING PROTOCOL INCLUSION CRITERIA:
* Patients must have histologically confirmed solid tumor requiring therapy and meet one of the following criteria:

  * Patients must have disease not amenable to curative-intent therapy OR
  * Patients who have had disease progression after treatment with all available therapies for their disease that are known to confer benefit or are intolerant to such treatment will be eligible, if other eligibility criteria are met. If the patient is currently receiving therapy without progression, the clinician must have assessed that the current therapy is no longer benefitting the patient, or that the patient is not tolerating the therapy. Patients can be screened on ADC MATCH if they are on first-line treatment and expected to need a treatment change within 3 months, and ADC MATCH is felt to be appropriate next line therapy OR
  * Patients with disease for which no standard treatment exists that has been shown to confer benefit OR
  * Patients who are willing to forego standard therapies known to confer benefit

    * NOTE: Patients can be on therapy at the time of initiating the Screening Protocol if the patient is interested in treatment on ADC MATCH upon progression, and the physician deems this appropriate
* Patient must have undergone RNA testing in a Clinical Laboratory Improvement Act (CLIA) environment. Patients who have high TOI RNA expression will have confirmation of TOI expression by CLIA IHC assay at MD Anderson Cancer Center (MDACC). Only patients with confirmed TOI protein expression will be eligible for assignment to a treatment cohort. Retrospective confirmation in another central laboratory may also be performed
* Patients must be willing to undergo mandatory pre-treatment and on-treatment tumor biopsies. Patients who do not consent to these research biopsies will not be eligible for prescreening. Patients who have screened and consented to a treatment cohort but are found to have disease that cannot be safely biopsied will be eligible for treatment provided all other eligibility criteria are met
* Patients must have measurable disease
* Age ≥ 18 years. Because no dosing or adverse event (AE) data are currently available on the use of the Cancer Therapy Evaluation Program (CTEP) investigational new drug (IND) agents to be used in the study in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group performance status of 0-2 (Karnofsky ≥ 50%)
* No history of transfusion dependence
* No history of persistent bone marrow suppression (absolute neutrophil count ≥ 1,500/mL and platelets ≥ 100,000/mL not attributable to active therapy; patients currently on bone marrow suppressive therapy can undergo assessment for the screening protocol but cannot be treated on any of the treatment cohorts unless bone marrow suppression is reversed off the suppressive therapy)
* Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN). Documented Gilbert syndrome is allowed if total bilirubin is ≤ 3 × ULN
* Aspartate transaminase (serum glutamic-oxaloacetic transaminase [SGOT])/alanine transaminase (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 × institutional ULN. Transaminases up to 5 × ULN in the presence of liver metastases are not allowed to initiate the screening protocol but are allowed for the treatment cohorts
* Creatinine ≤ institutional ULN OR glomerular filtration rate ≥ 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
* Patients must have albumin ≥ 3 g/dL
* Human immunodeficiency virus-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this study
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational agents are eligible for this study
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this study, patients should be class 2B or better
* Women of childbearing potential must have a negative human serum pregnancy test result at the screening protocol
* The effects of the study drugs on the developing human fetus are unknown. For this reason and because investigational agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after completion of study drug administration (unless otherwise indicated in the eligibility section of the treatment cohort protocols). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to study entry, for the duration of study participation, and for 6 months after completion of study drug administration
* Ability to understand and the willingness to sign a written informed consent document
* ADDITIONAL INCLUSION CRITERIA FOR TREATMENT COHORTS:
* Women of childbearing potential must have a negative serum pregnancy test result at treatment cohort screening
* Hemoglobin > 9.0 g/dL
* Leukocytes ≥ 3000/mL
* Absolute neutrophil count ≥ 1,500/mL
* Platelets ≥ 100,000/mL
* Patient must be willing to sign the relevant treatment cohort consent form
* COHORT A INCLUSION CRITERIA:
* Patients must fulfill all the eligibility criteria outlined in the ADC MATCH screening protocol at the time of treatment cohort A registration
* Patient must have high Trop-2 protein expression (IHC 2+ or 3+) as determined by the MD Anderson Cancer Center Clinical Laboratory Improvement Amendments IHC assay

  * Patients who have Trop-2 IHC testing without RNA testing or who have Trop-2 IHC 2 or 3+ expression but do not have Trop-2 expression detected on RNA testing will not be eligible for the trial.
  * Patients who have Trop-2 RNA expression and Trop-2 IHC 2+ or 3+ on another Trop-2 IHC test will undergo Trop-2 testing with the integral MDACC IHC assay
  * Patients who already have RNA expression testing demonstrating Trop-2 RNA expression as well as IHC testing on the MDACC CLIA lab platform will be eligible for enrollment after review of results by the Precision Oncology Decision Support team without having to repeat Trop-2 IHC results as part of pre-screening. Patients who have had TROP2 2+ testing result performed outside of MDACC will have to undergo MDACC TROP2 IHC analysis before enrollment
* COHORT B INCLUSION CRITERIA:
* Patients must fulfill all the eligibility criteria outlined in the ADC MATCH screening protocol at the time of treatment cohort B registration
* Patient must have high Nectin-4 protein expression (IHC 2+ or 3+) as determined by the MD Anderson Cancer Center Clinical Laboratory Improvement Amendments IHC assay
* COHORT C INCLUSION CRITERIA:
* Patients must fulfill all the eligibility criteria outlined in the ADC MATCH screening protocol at the time of treatment cohort C registration
* Patient must have HER2 protein expression (IHC 2+ or 3+) as determined by the MD Anderson Cancer Center (MDACC) IHC assay

  * Patients who have HER2 IHC testing without RNA testing or who have HER2 IHC 2 or 3+ expression but do not have HER2 expression detected on RNA testing will not be eligible for the trial
  * Patients who have HER2 RNA expression and HER2 IHC 3+ or 2+ on another HER2 IHC test will undergo HER2 testing with the integral MDACC IHC assay
  * Patients who already have RNA expression testing demonstrating HER2 RNA expression as well as IHC testing on the MDACC CLIA lab platform will be eligible for enrollment after review of results by the Precision Oncology Decision Support team without having to repeat HER2 IHC results as part of pre-screening. Patients who have had HER2 2+ testing result performed outside of MDACC will have to undergo MDACC HER2 IHC analysis before enrollment
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 7 months after completion of study drug administration. Women should not breastfeed during the study treatment period and for 7 months after completion of study drug administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to study entry, for the duration of study participation, and for 4 months after completion of study drug administration. Female patients must not donate, or retrieve for their own use, ova from the time of screening throughout the study treatment period and for at least 7 months after the final study drug administration. Female patients may wish to consider preservation of ova prior to enrollment in the study. Male patients should refrain from freezing or donating sperm during the study and for 6 months after the final study drug administration. Preservation of sperm should be considered prior to enrollment in the study
* LVEF ≥50% within 28 days before enrollment

Exclusion Criteria:

* SCREENING PROTOCOL EXCLUSION CRITERIA:
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease. Patients with treated brain metastases are eligible if follow-up brain imaging 4 weeks after central nervous system-directed therapy shows no evidence of progression
* Clinically significant cardiovascular condition including: (1) history of congestive heart failure (New York Health Association class > 2), (2) any history of unstable angina, (3) myocardial infraction within the past 12 months, or (4) any history of supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention
* History or presence of abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful
* Active or chronic corneal disorder including, but not limited to, Sjogren's syndrome, Fuchs corneal dystrophy (requiring treatment), history of corneal transplantation, active herpetic keratitis, and/or active ocular conditions requiring ongoing treatment/monitoring such as wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, presence of papilledema, and acquired monocular vision
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the ADCs used in the study
* History of interstitial lung disease or pneumonitis requiring steroid therapy
* Grade 2 or greater peripheral neuropathy
* Patients requiring the use of full dose coumarin-derivative anticoagulants such as warfarin. Low molecular weight heparin is permitted for prophylactic or therapeutic use. Factor X inhibitors are permitted

  * Note: Warfarin may not be started while enrolled in the treatment cohorts. Stopping the anticoagulation for biopsy should be per site standard operating practice
* Pregnant women are excluded from the study because the study drugs are investigational or approved agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with any of the study drugs, breastfeeding should be discontinued if the mother is treated with any of the study drug
* ADDITIONAL EXCLUSION CRITERIA FOR TREATMENT COHORTS:
* Patients must have adequate washout from prior therapy at the time of study treatment initiation: 4 weeks from major surgery; 4 weeks from antibody-based therapy; 2 weeks or 5 half-lives (whichever is shorter) from any targeted therapy or small molecule therapy; 3 weeks or 5 half-lives (whichever is shorter) from chemotherapy or 6 weeks in the case of certain therapies (e.g., extensive radiotherapy, mitomycin C, and nitrosoureas); and 4 weeks from radiation therapy. Patients should have received no more than 3 prior lines of chemotherapy. Testosterone suppression as supportive treatment for castration-resistant prostate cancer and ovarian suppression in premenopausal patients with breast cancer that have supportive treatment and not anticancer treatment role (with luteinizing hormone-releasing hormone analogs) will be allowed if the patients were on these supportive treatments before starting the study. Use of bone-modifying medications (bisphosphonates or denosumab) will be allowed. Palliative radiotherapy of non-target lesions is permitted, but presence of new or worsening metastases will be considered progressive disease. If there is clear evidence of clinical benefit, study treatment may be continued 2 weeks after completion of palliative radiotherapy to lesions that are non-target lesions. Patients can be on therapy during treatment cohort screening
* Patients who are currently receiving any other investigational agent(s)
* Received systemic therapy with corticosteroids at > 20 mg/day prednisone or equivalent within 1 week prior to cycle 1 day 1
* Patients who have not recovered from AEs due to prior anticancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* When the corrected QT interval (QTc) by Fridericia's formula is < 120 ms, > 450 ms in males and > 470 ms in females. When the QTc by Rautaharju's formula is ≥ 120 ms, > 450 ms in males and > 470 ms in females
* Uncontrolled infection requiring intravenous antibiotic, antiviral, or antifungal use
* Received a live, attenuated vaccine within 30 days prior to cycle 1 day 1. Enrolled patients should not receive live vaccine during the study. Non-live COVID vaccines will be allowed on study, but it is recommended to avoid their use during the first treatment cycle (from 3 days prior to cycle 1 day 1 through cycle 2 day 3)
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations
* COHORT A EXCLUSION CRITERIA:
* Patients with histologically documented advanced colorectal cancer, urothelial cancer, head and neck cancer, triple negative breast cancer (TNBC), HR-positive breast cancer, HER2-positive breast cancer, small cell lung cancer, NSCLC, and endometrial cancer
* Patients who have received growth factor support within 2 weeks of study treatment initiation
* Coadministration of sacituzumab govitecan (IMMU-132) with inhibitors of UGT1A1 may increase systemic exposure to the active metabolite, SN-38. UGT1A1 inhibitors should not be administered concomitantly with sacituzumab govitecan (IMMU-132) unless there are no therapeutic alternatives
* Prior topoisomerase 1 inhibitor treatment
* Prior treatment with a Trop-2-targeting ADC
* Has active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal (GI) perforation within 6 months of treatment cohort A registration
* COHORT B EXCLUSION CRITERIA:
* Patients with histologically documented advanced urothelial cancer, head and neck cancer, breast cancer, lung cancer, gastric cancer, gastroesophageal junction cancer, esophageal cancer, prostate cancer, or penile cancer
* Concomitant use of strong inhibitors or strong inducers of cytochrome P450 (CYP)3A4. Washout period is 2 weeks prior to study treatment initiation
* History of uncontrolled diabetes mellitus within 3 months before the first dose of study treatment. Uncontrolled diabetes mellitus is defined as hemoglobin A1c ≥ 8% or hemoglobin A1c between 7 and < 8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained
* Known active keratitis or corneal ulcerations. Patients with superficial punctate keratitis are allowed if the disorder is being adequately treated
* Known hypersensitivity to enfortumab vedotin or to any excipient in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate, and polysorbate 20), or known hypersensitivity to biopharmaceutical produced in Chinese hamster ovary cells
* Prior treatment with an ADC with vedotin payload
* COHORT C EXCLUSION CRITERIA:
* Patients with histologically documented advanced breast cancer, non-small cell lung cancer (NSCLC), colorectal carcinoma (CRC), gastric cancer, or gastroesophageal junction (GEJ) cancer
* Previous treatment with topoisomerase I inhibitors as a free form or as other formulations, and ADCs with topoisomerase I inhibitor payloads
* Patients receiving treatment with chloroquine or hydroxychloroquine are not allowed to participate in the study, unless there is a washout period of at least 14 days prior to the first dose of study drug
* History of non-infectious pneumonitis/interstitial lung disease (ILD), current ILD, or where suspected ILD that cannot be ruled out by imaging at screening
* Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (i.e., pulmonary emboli within 3 months of initiation of study drug, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion etc.)
* Any autoimmune, connective tissue or inflammatory disorders (e.g., Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening
* Prior pneumonectomy
* History of severe hypersensitivity reactions to other monoclonal antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of high protein expression in patients with high ribonucleic acid (RNA) expression of each antibody-drug conjugate target (screening protocol) | Up to completion of screening period
Objective response rate (treatment cohorts) | Up to 3 years
  Will be defined as the proportion of patients who achieve complete response or partial response per the Response Evaluation Criteria in Solid Tumors version 1.1. For each treatment cohort, 90% two-sided confidence intervals will be calculated for objective response rate.

SECONDARY OUTCOMES:
Frequency that patients with high RNA and immunohistochemistry target expression receive cohort treatment on study (screening protocol) | Up to 3 years
Progression free survival (treatment cohorts) | From start of cohort treatment to time of progression or death, assessed at 6 months
  Will be estimated using the Kaplan-Meier method. For each treatment cohort, 90% two-sided confidence intervals will be calculated for the proportion of patients alive and progression free at 6 months from start of cohort treatment.
Overall survival (treatment cohorts) | From start of cohort treatment to time of death, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method.
Time to progression (treatment cohorts) | Up to 3 years
  Will be estimated using the Kaplan-Meier method.
Incidence of adverse events (treatment cohorts) | Up to 30 days after completion of study treatment
  Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
RNA expression of targets of interest (TOIs) (treatment cohorts) | Up to 3 years
  Pearson and Spearman correlation will be calculated to assess the correlation of RNA and protein expression of TOIs.
Temporal tumor heterogeneity (treatment cohorts) | Up to 3 years
  Paired t-test will be used to determine temporal tumor heterogeneity by comparing RNA/protein expression of TOIs on archival samples versus fresh biopsies. Graphic methods will be used to depict the temporal changes in RNA/protein expression of TOIs over time.
Potential predictive biomarkers and other molecular features (treatment cohorts) | Up to 3 years
  Logistic regression (or chi-squared test) or proportional hazard model (or log-rank test) will be used to identify potential predictive biomarkers, including target expression and other molecular features, for predicting response endpoints or survival endpoints.
Pharmacodynamic changes in the tumor and microenvironment (treatment cohorts) | Up to 3 years

OTHER OUTCOMES:
Mechanisms of acquired resistance (treatment cohorts) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (26):
- United States (26):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm